CLINICAL TRIAL: NCT07347288
Title: An Open-label, Multicenter Exploratory Clinical Study of the EZH2 Inhibitor SHR2554 as Maintenance Therapy After First-line Systemic Treatment in Patients With Peripheral T-cell Lymphoma
Brief Title: SHR2554 as Maintenance Therapy in Patients With Peripheral T-cell Lymphoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-SR-1121
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: PTCL

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR2554 monotherapy (Experimental): Patients With Peripheral T-cell Lymphoma After First-line Systemic Treatment Receiving SHR2554 monotherapy as Maintenance Therapy
  Interventions: Drug: SHR2554 Tablets

INTERVENTIONS:
Drug: SHR2554 Tablets — SHR2554 orally twice daily

SUMMARY:
Evaluation of the Safety and Efficacy of SHR2554 as Maintenance Therapy after first-line systemic treatment in patients with peripheral T-cell lymphoma

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Histologically confirmed PTCL,including PTCL NOS, ALCL, nTFHL,MEITL,ENKTL etc. according to WHO 2022 criteria.
3. Previously received first-line systemic induction therapy and achieved CR/PR; Auto-transplantation or allo-transplantation are allowed.
4. A measurable or evaluable disease at the time of first diagnosis of PTCL (any nodes/nodal masses>1.5 cm in longest diameter (LDi) or extralymphatic sites of disease >1.0 cm in LDi)
5. ECOG PS 0-2
6. With adequate organ function
7. Expected survival ≥ 12 weeks
8. Women of childbearing potential (WOCBP) should be proven to be negative by human chorionic gonadotropin (hCG) test in 7 days before the first dose of SHR2554. They must be willing and able to employ a highly effective method of birth control/contraception to prevent pregnancy from the day they sign the informed consent form (ICF) to at least 30 days after receiving the last dose of study treatment. Male subjects with WOCBP partner should receive Surgical sterilization or consent to employ a highly effective method of birth control/contraception to prevent pregnancy；
9. Participant who has provided written consent to participate in the study and ability to comply with all aspects of the protocol.

Exclusion Criteria:

1. cutaneous T cell lymphoma
2. Has a prior malignancy other than the malignancies under study within 3 years without relieve
3. Participants with a presence of central nerves invasion
4. Known sensitivity or allergy to investigational product
5. Participated in another clinical trial within 4 weeks prior to the start of the study;
6. Women who are pregnant or lactating. Patients have breeding intent in 12 months or cannot take effective contraceptive measures during the trial measures
7. Active infected persons, except tumor-related B symptom fever;
8. Diseases and medical history:

1.have multiple factors that affect oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction); 2.have a history of psychotropic substance abuse and can not quit or have mental disorders; 3.Subjects with any severe and/or uncontrolled medical condition; 9.A history of immunodeficiency 10.Patients with mental disorders or those unable to provide informed consent 11.In any conditions which investigator considered ineligible for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
2 years PFS | 2 years
  The 2-year rate of during and after treatment that the participant lives without progression of the disease, as assessed by 2014 Lugano criteria.

SECONDARY OUTCOMES:
1-year and 2-year DFS rates for patients who were in CR at enrollment | 1year,2year
  The rate of 1-year and 2-year that the participant lives without disease, as assessed by 2014 Lugano criteria.
Rate of patients who were PR at enrollment converting to CR | Time from the first dose to any events, assessed up to 12 months
  The Rate of patients who were PR at enrollment converting to CR
Complete Response Rate (CR) | Time from the first dose to disease progression or death, assessed up to 12months
  The proportion of participants who achieve a complete response (CR) during the treatment period, as assessed by the 2014 Lugano criteria using FDG-PET imaging.
Duration of Response (DoR) | From the date response is first documented to the date of disease progression or death, up to 36 months
  The interval from the initial documentation of response (CR or PR) to the first documentation of disease progression or death.
Progression-Free Survival (PFS) | Time from the first dose to disease progression or death, assessed up to 36 months
  The length of time during and after treatment that the participant lives without progression of the disease, as assessed by 2014 Lugano criteria.
Overall Survival (OS) | Time from the first dose to death from any cause, assessed up to 36 months
  The length of time from the start of treatment until death from any cause.
Incidence of Treatment-Related Adverse Events (Safety and Tolerability) | Up to 12 months
  The incidence, type, and severity of adverse events (graded according to CTCAE v5.0), and their relationship to the study treatment.

OTHER OUTCOMES:
Minimal Residual Disease (MRD)-Negative Rate | Up to 12 months after the first dose
  The proportion of patients who achieve minimal residual disease negativity at the completion of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes